CLINICAL TRIAL: NCT01139476
Title: Study of Biomarkers of Exposure and Effects in Agriculture
Brief Title: Specimen Collection for Agricultural Health Study Cohort Pesticide Exposure Study
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999910106; 10-C-N106
Record Dates: First submitted 2010-06-05; First posted 2010-06-08 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-04-18

CONDITIONS: Multiple Myeloma; Leukemia; MGUS; Monoclonal B-Cell Lymphocytosis
Keywords: Multiple Myeloma; MGUS; Leukemia; Biorepository; Natural History
MeSH Terms: conditions — Multiple Myeloma; Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AHS BEEA participants: A subset of 1990 AHS cohort members who are male private pesticide applicators, living and over 50 years of age at the time contact, cancer free, and who completed AHS Phases IIII.
- Non-AHS BEEA participants: A group of 225 age-, race-, and countymatched, non-AHS controls, who have not lived or worked on a farm as an adult, or held a job applying pesticides.

SUMMARY:
Background:

- Multiple myeloma (MM), a type of cancer that affects the white blood cells, is often preceded by a precancerous disorder known as monoclonal gammopathy of undetermined significance (MGUS). Farmers and other agricultural workers have a higher risk of developing MGUS and MM, possibly because of their exposure to certain pesticides. Researchers are interested in studying biological specimens taken from participants in the Agricultural Health Study - specifically, pesticide applicators at least 50 years of age who do not have cancer- to better understand the development of MGUS and MM.

Objectives:

* To collect biological specimens from Agricultural Health Study participants for further research.
* To examine the relationship between pesticide exposure and MGUS/MM.

Eligibility:

- Male pesticide applicators who are over 50 years of age, cancer-free, and participating in the Agricultural Health Study.

Design:

* Two groups of participants will complete the study: a general group and a smaller group of individuals who have been exposed to the pesticide diazinon.
* All participants will receive an initial contact letter with information about the study, followed by a phone call to administer a screening questionnaire and arrange a home visit from a researcher within the next month.
* Participants will receive by mail a urine specimen kit that will be collected at the home visit.
* During the home visit, a study researcher will take blood samples and collect the urine sample, and will administer another questionnaire.
* Participants in the group exposed to diazinon will have three home visits for the study: (1) prior to pesticide exposure, (2) the day after participants stop using diazinon, and (3) about 21 days after the second visit. The first visit will take place in the off-season from January to March; the second and third visits will be conducted between April and August.
* No treatment will be provided as part of this study.

DETAILED DESCRIPTION:
We propose to conduct a molecular epidemiology study with a subset of participants in the Agricultural Health Study (AHS), a prospective cohort of 57,310 licensed pesticide applicators in Iowa and North Carolina. Blood and urine samples will be collected from 1,990 cancer-free male AHS participants over the age of 50. These participants will also be asked to complete a brief interview (approximately 20 minutes) regarding recent exposures and other lifestyle and health characteristics, which will be conducted at the time of the biospecimen collection. Participants in both Iowa and North Carolina will be enrolled and home visits for interviews and sample collection will take place throughout the year between 2010-2014.

The proposed study has two primary objectives. First, we will determine the prevalence and study the etiology of monoclonal gammopathy of undetermined significance (MGUS), which is a precursor biomarker for multiple myeloma. We will compare the prevalence of MGUS in the AHS cohort with the prevalence in two general population-based cohorts ( i.e., Olmsted County and NHANES IID) with well-characterized MGUS prevalence levels. As a result of previous data collection efforts in the AHS, comprehensive information on lifetime occupational exposures and lifestyle factors will be available for the subjects included in this study. We will examine the associations between MGUS and lifetime exposure to specific pesticides within the AHS cohort. We will also evaluate several other biomarkers, including telomere length and global DNA hypomethylation in peripheral blood lymphocytes, for associations with specific pesticides and excess risk of MGUS.

The second objective is to establish a resource with the remaining blood and urine samples collected from the participants in this study. These biospecimens will be used to evaluate the biological plausibility and the mechanism-of-action of associations between pesticides and cancers observed in earlier AHS studies. Many of these pesticides are non-genotoxic and their mechanism of carcinogenesis has not been determined. One such future study involving repository samples will be an investigation of monoclonal B-cell lymphocytosis (MBL), a marker which has been shown to precede chronic lymphocytic leukemia in previous studies. Several pesticides in current widespread use in the AHS have been linked to leukemia. We will determine the prevalence of MBL in the AHS cohort and evaluate potential associations with specific pesticides of interest to better explain the relation between pesticide exposures and leukemia risk.

ELIGIBILITY:
* INCLUSION CRITERIA:

Selected participants in the Agricultural Health Study are invited to participate in this aspect of the study.

1. Male private pesticide applicator;
2. Alive as of the latest update of the National Death Index G\fDD and over 50 years of age at the time of initial contact:
3. Cancer free as of the most recent linkage with the appropriateCancer Registry;
4. Completed phase I, II and III interviews (these study subjects have the most comprehensive exposure evaluation and also will be the most interested in the study).

EXCLUSION CRITERIA:

1. Deceased or no longer residing in Iowa or North Carolina;
2. Ever diagnosed with any type of cancer other than non-melanoma skin cancer;
3. Unable to speak English;
4. Have a blood clotting disorder such as hemophilia; or
5. Registered with the AHS as a "no contact".

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male pesticide applicators who are over 50 years of age, cancer-free, and participating in the Agricultural Health Study. Plus, a small control group comprising individuals who have not worked in agriculture or been occupationally exposed to pesticides.
Sampling Method: Non-Probability Sample
Enrollment: 1892 (Actual)
Dates: Start 2010-06-15

PRIMARY OUTCOMES:
No intervention; looking for associations between MGUS and specific pesticides within the AHS cohort and whether selected biomarkers are associated with excess MGUS | Most participants receive specimen collection at one time-point (home visit); selected participants receive specimen collection at three time-points (home-visit)
  To collect biological specimens from Agricultural Health Study participants for further research. To examine the relationship between pesticide exposure and MGUS/MM.

SECONDARY OUTCOMES:
Establish a resource with the remaining biospecimens collected from the participants of the MGUS study that will be used to evaluate the biological plausibility and the mechanism-of-action of associations between pesticides and cancers in earlie... | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan N Hofmann, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- University of Iowa, Iowa City, Iowa, United States